CLINICAL TRIAL: NCT02493270
Title: Effect of Smoking Cessation on Non-surgical Periodontal Therapy
Acronym: EsCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Claudio Mendes Pannuti, Associate Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EsCAPE
Record Dates: First submitted 2015-07-02; First posted 2015-07-09 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Periodontitis
Keywords: smoking cessation; tobacco; dental; periodontal
MeSH Terms: conditions — Periodontitis; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adjunctive smoking cessation (Experimental): non-surgical periodontal therapy and concurrent smoking cessation therapy
  Interventions: Behavioral: Smoking cessation therapy; Procedure: Non-surgical periodontal therapy

INTERVENTIONS:
Behavioral: Smoking cessation therapy — Multidisciplinary smoking cessation therapy, performed by a team comprising physicians, nurses, a psychologist and dentists. It consisted of four 1-h counselling lectures, psychologist-assisted cognitive behavioural therapy, nicotine replacement therapy and medication (bupropion or varenicline). Smoking cessation motivation was reinforced by dentists at the maintenance sessions, by means of motivational interviewing techniques
Procedure: Non-surgical periodontal therapy — full-mouth supra and subgingival scaling and root planing (with curettes and ultrasonic scaler); oral hygiene instruction and motivation and removal of intra-oral plaque retentive factors

SUMMARY:
The aim of this prospective study is to verify the efficacy of smoking cessation on non-surgical periodontal therapy in adult subjects with chronic periodontitis.

Smokers that were willing to quit received periodontal treatment and concurrent smoking cessation therapy. Periodontal maintenance was performed every 3 months. A calibrated examiner, blinded to smoking status, assessed periodontal status, gathered demographic and behavioural information with a structured questionnaire and measured air carbon monoxide concentration measurements.

ELIGIBILITY:
Inclusion Criteria:

* subjects were willing to stop smoking
* >10 teeth
* periodontitis (30% or more of their teeth with proximal CAL ≥ 5 mm

Exclusion Criteria:

* systemic conditions considered as risk factors for periodontal disease,
* periodontal therapy in the last 6 months
* continuous systemic use of anti-inflammatory or steroidal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2007-05; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Attachment Level (millimeters) after 24 months | baseline and 24 months

SECONDARY OUTCOMES:
Change in Gingival recession (millimeters) after 24 months | baseline and 24 months
Change in Pocket depth (millimeters) after 24 months | baseline and 24 months
Change in bleeding on probing (percentage of sites with bleeding) after 24 months | baseline and 24 months
Change in visible plaque (percentage of sites with visible plaque) after 24 months | baseline and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudio M Pannuti, PhD, Principal Investigator — University of Sao Paulo

REFERENCES:
- [Result] Rosa EF, Corraini P, Inoue G, Gomes EF, Guglielmetti MR, Sanda SR, Lotufo JP, Romito GA, Pannuti CM. Effect of smoking cessation on non-surgical periodontal therapy: results after 24 months. J Clin Periodontol. 2014 Dec;41(12):1145-53. doi: 10.1111/jcpe.12313. Epub 2014 Nov 21. PMID 25265872
- [Result] Rosa EF, Corraini P, de Carvalho VF, Inoue G, Gomes EF, Lotufo JP, De Micheli G, Pannuti CM. A prospective 12-month study of the effect of smoking cessation on periodontal clinical parameters. J Clin Periodontol. 2011 Jun;38(6):562-71. doi: 10.1111/j.1600-051X.2011.01723.x. Epub 2011 Apr 13. PMID 21488933